CLINICAL TRIAL: NCT05812209
Title: Stellate Ganglion Block to Treat Long COVID-19 Syndrome, A 41 Patient Retrospective Cohort Study
Brief Title: Stellate Ganglion Block to Treat Long COVID 19 Case Series
Status: Completed | Type: Observational
Sponsor: Metamorphosis LTD (Other)
Responsible Party: Principal Investigator, Lisa Pearson, Dr. Lisa Pearson, CRNA, NSPMc, Metamorphosis LTD
Other Study IDs: SGBCOVID
Record Dates: First submitted 2023-04-10; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Long COVID; Long Covid19; Post-COVID-19 Syndrome; Post Acute COVID-19 Syndrome; Dysautonomia; Anosmia; Dysgeusia; Brain Fog; Muscle Pain; Shortness of Breath; Dizziness; Fatigue Post Viral; Cough; Menstrual Cycle Abnormal; Pain
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Autonomic Nervous System Diseases; Anosmia; Dysgeusia; Mental Fatigue; Myalgia; Dyspnea; Dizziness; Cough; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SGB Patients for Long COVID 19: Patients who received ultrasound guided Stellate Ganglion block for symptoms of Long COVID in our Colorado clinics.
  Interventions: Procedure: Stellate Ganglion Block

INTERVENTIONS:
Procedure: Stellate Ganglion Block — Ultrasound guided block of the Stellate Ganglion with local anesthetics.
  Other Names: SGB

SUMMARY:
An assessment of the effectiveness of Stellate Ganglion Block in alleviating symptoms of Long COVID-19.

DETAILED DESCRIPTION:
We evaluated the treatment results of 41 patients (18 male and 23 female) aged between 18 and 89, who received Stellate Ganglion Block (SGB) with Ultrasound guidance for Long COVID-19 Syndrome. The patients were from the United States and received treatment at our Colorado clinics during the period of September to December 2022.Those who responded to our post-procedure follow-up calls were included in the study population.

ELIGIBILITY:
Inclusion Criteria: People who scheduled themselves for a SGB in our clinics in Colorado.

-

Exclusion Criteria:

Stellate Ganglion Block Contraindications

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study included 18 male and 23 females with an age range between 18 and 89 who underwent stellate ganglion block (SGB) for long COVID-19 Syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Symptom Response | 3 months
  Evaluation of the symptoms response to the Stellate Ganglion Block

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Pearson, DNAP, Principal Investigator — Metamorphosis LTD
Locations (1):
- Metamorphosis LTD, Cañon City, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan to share data file
Supporting Information: SAP, CSR
Time Frame: Within a month